CLINICAL TRIAL: NCT01985477
Title: Phase I/II Study of Lenalidomide (Revlimid), All-trans Retinoic Acid (ATRA) and Dexamethasone in Patients With Relapsed/Refractory Multiple Myeloma
Brief Title: Revlimid / All-Trans Retinoic Acid (ATRA) / Dexamethasone in Relapsed/Refractory Multiple Myeloma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Terminated Phase I due to slow accrual without progression to Phase II.
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2013-0624; NCI-2014-01098 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2013-11-08; First posted 2013-11-15 (Estimated); Last update posted 2016-09-14 (Estimated); Status verified 2016-09

CONDITIONS: Myeloma
Keywords: Myeloma; Multiple myeloma; MM; Relapsed/Refractory Multiple Myeloma; RR MM; Lenalidomide; CC-5013; Revlimid; Dexamethasone; Decadron; All-Trans Retinoic Acid; ATRA; Tretinoin (Oral); Vesanoid
MeSH Terms: conditions — Neoplasms, Plasma Cell; Multiple Myeloma | interventions — Lenalidomide; Dexamethasone; Calcium Dobesilate; Tretinoin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lenalidomide + Dexamethasone + All-Trans Retinoic Acid (ATRA) (Experimental): Phase I All Patients - Induction: Lenalidomide starting dose 25 mg by mouth 1 time every day on Day 1-21. Dexamethasone starting dose 40 mg by mouth on Days 1,8,15,22. ATRA starting dose 25 mg/m2 by mouth 2 times each day on Days 1-21.
  Phase II Group A: Lenalidomide starting dose: Dose tolerated prior to enrollment. Dexamethasone starting dose: Dose previously on when progressing prior to study entry. ATRA starting dose: MTD from Phase I.
  Maintenance Therapy Group A: Lenalidomide at dose level tolerated at completion of cycle 3 for 21/28 days, with ATRA at dose determined in Phase I for 14/28 days, and Dexamethasone at last tolerated dose on Days 1, 8, 15 and 22. After 3 months on therapy at MTD in Phase I study, patients must be switched to this dose schedule. Patients unable to tolerate either Dexamethasone during maintenance phase may dose reduce Dexamethasone as needed.
  Interventions: Drug: Lenalidomide; Drug: Dexamethasone; Drug: All-Trans Retinoic Acid (ATRA)
- Lenalidomide + All-Trans Retinoic Acid (ATRA) (Experimental): Phase II Group B: Lenalidomide will be given as a single oral dose at the level patient was on at the time of progression on single agent Lenalidomide prior to study enrollment. All-Trans Retinoic Acid (ATRA) starting dose: MTD from Phase I.
  Maintenance Therapy: Maintenance therapy consists of lenalidomide at the dose level tolerated at the completion of cycle 3 for 21/28 days, with ATRA at the dose determined in the phase I portion of the trial for 14/28 days. Dexamethasone will not be administered. After 3 months on therapy at the MTD in the phase 1 study, patients must be switched to this dose schedule.
  Interventions: Drug: Lenalidomide; Drug: All-Trans Retinoic Acid (ATRA)

INTERVENTIONS:
Drug: Lenalidomide — Phase I All Patients - Induction: Lenalidomide starting dose 25 mg by mouth 1 time every day on Day 1-21.
  Phase II Group A: Lenalidomide starting dose: Dose tolerated prior to enrollment.
  Maintenance Therapy: Phase I and Phase II Group A: Maintenance therapy lenalidomide at dose level tolerated at completion of cycle 3 for 21/28 days.
  Phase II Group B: Lenalidomide will be given as a single oral dose at the level patient was on at the time of progression on single agent lenalidomide prior to study enrollment.
  Other Names: CC-5013; Revlimid
Drug: Dexamethasone — Phase I All Patients - Induction: Dexamethasone starting dose 40 mg by mouth on Days 1,8,15,22.
  Phase II Group A: Dexamethasone starting dose: Dose previously on when progressing prior to study entry.
  Maintenance Therapy: Phase I and Phase II Group A: Dexamethasone at last tolerated dose on Days 1, 8, 15 and 22.
  Other Names: Decadron
  Arms: Lenalidomide + Dexamethasone + All-Trans Retinoic Acid (ATRA)
Drug: All-Trans Retinoic Acid (ATRA) — Phase I All Patients - Induction: ATRA starting dose 25 mg/m2 by mouth 2 times each day on Days 1-21.
  Phase II Group A: ATRA starting dose: MTD from Phase I.
  Maintenance Therapy: Phase I and Phase II Group A: ATRA at dose determined in Phase I for 14/28 days.
  Phase II Group B: All-Trans Retinoic Acid (ATRA) starting dose: MTD from Phase I.
  Maintenance Therapy Group B: ATRA at the dose determined in the Phase I portion of the trial for 14/28 days.
  Other Names: ATRA; Tretinoin (Oral); Vesanoid

SUMMARY:
The goal of the Phase I portion of this clinical research study is to find the highest tolerated dose of the combination of lenalidomide, all-trans retinoic acid (ATRA), and dexamethasone that can be given to patients with relapsed or refractory multiple myeloma (MM).

The goal of the Phase II portion of this study is to learn if ATRA when given in combination with lenalidomide alone or with lenalidomide and dexamethasone can help to control multiple myeloma.

In September 2015, the study was terminated due to slow accrual while still a Phase I study, no additional registration or research performed under the Phase II portion of the study.

DETAILED DESCRIPTION:
Study Groups:

If you are found to be eligible to take part in this study, you will be assigned to a study group based on when you joined this study. Up to 2 groups of up to 3-6 patients participants will be enrolled in the Phase I portion of the study, and up to 58 participants will be enrolled in Phase II.

If you are enrolled in the Phase I portion, the dose of lenalidomide, dexamethasone, and ATRA you receive will depend on when you joined this study. The first group of participants will receive the lowest dose level of the combination. Each new group will receive a higher dose of the combination than the group before it, if no intolerable side effects were seen. This will continue until the highest tolerable dose of the combination of lenalidomide and ATRA is found.

If you are enrolled in the Phase II portion, you will be assigned to 1 of 2 groups based on the therapy you were receiving before you began to take part in this study.

* If you were receiving lenalidomide alone, you will take lenalidomide and ATRA (Group A).
* If you were receiving lenalidomide and dexamethasone when you started this study, you will take lenalidomide, dexamethasone, and ATRA (Group B).

Study Drug Administration:

Each cycle is 28 days.

The first part of the study, called induction, will have 3 cycles. After that is the maintenance part of the study. You will be able to continue on maintenance for as long as the doctor thinks it is in your best interest.

Induction:

* On Day 1-21 of each cycle, you will take lenalidomide by mouth 1 time every day.
* On Days 1-21 of each cycle, you will take ATRA by mouth 2 times each day.
* On Days 1, 8, 15, and 22 of each cycle (+/- 3 days), you will take dexamethasone by mouth.

Maintenance:

* On Day 1-21 of each cycle, you will take lenalidomide by mouth 1 time every day.
* On Days 1-14 of each cycle, you will take ATRA by mouth 2 times each day.
* If you are in Group A, on Days 1, 8, 15, and 22 of each cycle (+/- 3 days), you will take dexamethasone by mouth.

If a dose of lenalidomide is missed or vomited, you should continue with the regular schedule of the drug at the next dose, and a missed dose should NOT be made up.

Lenalidomide capsules should be swallowed whole, and should not be broken, chewed or opened. If you take more than the prescribed dose of lenalidomide, you should seek emergency medical care if needed and contact study staff right away

Study Visits:

Induction Study Visits:

On Days 1, 8, and 15 of Cycle 1:

* You will have a physical exam.
* Blood (about 3 tablespoon) will be drawn for routine tests.
* Urine will be collected over 24 hours to check the status of the disease (Day 1 only).

Between Days 19 and 21 of Cycle 1, you will have a bone marrow aspiration and blood (about 1 teaspoon) will be drawn to measure the levels of certain proteins for research purposes.

On about Day 1 of Cycles 2-3:

* You will have a physical exam.
* Blood (about 3 tablespoons) will be drawn for routine tests
* Blood (about 1 teaspoon) will be drawn to measure proteins in your blood.
* Urine will be collected over 24 hours to check the status of the disease.

If your doctor thinks it is needed, the visits may take place more often. You may have extra visits at any time during the study if your doctor thinks it is needed for your care.

Maintenance Therapy Study Visits:

Once a month during Maintenance Therapy:

* You will have a physical exam.
* Blood (about 2 teaspoons) will be drawn for routine tests.
* Blood (about 1 teaspoon) will be drawn to measure proteins in your blood.
* Urine will be collected over 24 hours to check the status of the disease.
* If the doctor thinks it is needed, you will have a bone marrow biopsy to check the status of the disease.

Length of Study:

You will receive up to 3 cycles of the study drugs during induction. You may continue taking the study drugs during maintenance for as long as the doctor thinks it is in your best interest. You will no longer be able to take the study drug if the disease gets worse if intolerable side effects occur, or you are unable to follow study directions.

Your participation on this study will be over after the end-of-study visit.

End-of-Study Visit:

If you go off study for any reason, you will have an end-of-study visit. This is usually done about 30 days after the last dose of the study drugs. At this visit, the following tests and procedures will be performed:

* You will have a physical exam.
* Blood (about 2-3 teaspoons) and urine (over 24 hours) will be collected to check the status of the disease.
* Blood (about 1 tablespoon) will be drawn for routine tests.
* If the doctor thinks it is needed, you will have a bone marrow biopsy to check the status of the disease.

This is an investigational study. ATRA is FDA approved and commercially available to treat acute promyelocytic leukemia.

Lenalidomide is FDA approved and commercially available to treat MM.

Dexamethasone is FDA approved and commercially available to treat inflammation and allergic conditions and to manage the symptoms of several types of leukemia and lymphoma.

The combination of ATRA, lenalidomide, and dexamethasone is investigational.

Up to 70 participants will be enrolled in this study. All will take part at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Understand and voluntarily sign an informed consent form
2. Age >/= 18 years at the time of signing the informed consent form
3. Serum creatinine </= 2.5 mg/dl OR Creatine clearance > 30 ml/min
4. Eastern Cooperative Oncology Group (ECOG) performance status score of 0, 1, or 2
5. Females of childbearing potential (FCBP)* must have a negative serum or urine pregnancy test with a sensitivity of at least 50 mlU/mL within 10-14 days prior to and again within 24 hours of starting lenalidomide and must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional affective method AT THE SAME TIME, at least 28 days before she starts taking lenalidomide. FCBP must also agree to ongoing pregnancy testing. Men must agree to use a latex condom during sexual contact with a female of childbearing potential even if they have had a successful vasectomy. All patients must be counseled at a minimum of every 28 days about pregnancy precautions and risks of fetal exposure.
6. Continuation from Inclusion #5: *A female of childbearing potential is a sexually mature woman who: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months).
7. Able to take prophylactic antiplatelet/anticoagulation, warfarin or equivalent agent
8. Patient is able to understand and comply with the terms and conditions of the Lenalidomide Counseling Program.
9. Phase I Specific Inclusion Criteria: Multiple myeloma that has progressed on lenalidomide and dexamethasone combination therapy at a dose of 25 mg daily on lenalidomide and 40 mg weekly of dexamethasone with measurable levels of myeloma paraprotein in serum ( >/= 0.5 g/dl), urine ( >/= 0.2 g excreted in a 24-hour collection sample), or abnormal free light chain (FLC) ratio.
10. Phase I Specific Inclusion Criteria: Laboratory test results within these ranges: Absolute neutrophil count > 1000 cells/mm^3; Platelet count > 100,000 cells/mm^3 for patients with < 50% of bone marrow plasma cells and platelet count > 50,000 cells/mm^3 for patients in whom > 50% of the bone marrow nucleated cells were plasma cells; Total bilirubin </= 2.0 mg/dL; AST (SGOT) and ALT (AGPT) < 3 x upper limits of normal (ULN)
11. Phase II Specific Inclusion Criteria: Cohort A: Multiple myeloma that has progressed on lenalidomide and dexamethasone combination therapy with measurable levels of myeloma paraprotein in serum ( >/= 0.5 g/dl), urine ( >/= 0.2 g excreted in a 24-hour collection sample), or involved FLC level by more than 10 mg/dL and abnormal free light chain (FLC) ratio. Cohort B: Multiple myeloma that has progressed on single agent lenalidomide therapy with measurable disease defined as: doubling of the M-component in 2 consecutive measurements in less than or equal to 2 months OR increase in serum M-protein levels by >/= .5g or urine protein by 200mg/24 hours, or involved FLC level by more than 10 mg/dL (with an abnormal FLC ratio).
12. Phase II Specific Inclusion Criteria: Laboratory test results within these ranges: Absolute neutrophil count > 1000 cells/mm^3; Platelet count > 75,000 cells/mm^3 for patients with < 50% of bone marrow plasma cells and platelet count > 50,000 cells/mm^3 for patients in whom > 50% of the bone marrow nucleated cells were plasma cells; Total bilirubin </= 2.0 mg/dL; AST (SGOT) and ALT (AGPT) < 3 x ULN

Exclusion Criteria:

1. Any serious medical condition, or psychiatric illness that would prevent the subject from signing the informed consent form.
2. Pregnant or breast feeding females. (Lactating females must agree not to breast feed while taking lenalidomide).
3. Use of any cancer therapy within 14 days prior to beginning cycle 1 day 1 of therapy with the exception of lenalidomide and dexamethasone (radiation therapy allowed within 5 days of completion of radiation therapy)
4. Known hypersensitivity to lenalidomide or ATRA.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2013-12; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of Lenalidomide/Dexamethasone and All-Trans Retinoic Acid (ATRA) | 28 days
  MTD defined as highest dose level in which 6 patients have been treated with less than 2 instances of dose limiting toxicity (DLT). Dose limiting toxicity refers to a medically significant event which meets one of the following:
  Hematologic dose-limiting toxicity defined as either, Grade 4 neutropenia lasting for >/=14 days in duration ( growth factors permitted after DLT established), Grade 4 thrombocytopenia > 14 days despite platelet transfusions.
  Non-hematologic DLT defined as any Grade 3, 4 or 5 non-hematologic toxicity, with the specific exception of, Isolated Grade 3 elevation of liver function tests (LFTs) without associated clinical symptoms, lasting for </=7 days in duration, Isolated Grade 3 elevation of amylase without associated clinical symptoms, Grade 3 hypocalcemia, hyperglycemia, hypokalemia, hypomagnesemia, hyponatremia, or hypophosphatemia which responds to medical intervention.

SECONDARY OUTCOMES:
Objective Response | After 4, 28 day cycles
  The objective response (complete response + partial response) at 4 cycles is the primary endpoint. Patients assessed for response each cycle of therapy according to International Myeloma Working Group Criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Jatin J. Shah, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org